CLINICAL TRIAL: NCT05582395
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate Mavacamten in Adults With Symptomatic Non-obstructive Hypertrophic Cardiomyopathy
Brief Title: A Study of Mavacamten in Non-Obstructive Hypertrophic Cardiomyopathy
Acronym: ODYSSEY-HCM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV027-031; U1111-1269-8581 (Registry Identifier: WHO); 2023-506352-24 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-09-14; First posted 2022-10-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: Mavacamten; non-obstructive HCM; non-obstructive hypertrophic cardiomyopathy (nHCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mavacamten (Experimental)
  Interventions: Drug: Mavacamten
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mavacamten — Specified dose on specified days
  Other Names: BMS-986427; MYK-461
  Arms: Mavacamten
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of mavacamten compared with placebo in participants with symptomatic non-obstructive hypertrophic cardiomyopathy (nHCM).

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of HCM consistent with current American College of Cardiology Foundation/American Heart Association and European Society of Cardiology guidelines: unexplained left-ventricular hypertrophy with non-dilated ventricular chambers in the absence of other cardiac or systemic disease which can produce the required magnitude of hypertrophy of a maximal left ventricular (LV) wall thickness ≥ 15 millimeters (mm) (or ≥ 13 mm with positive family history of hypertrophic cardiomyopathy [HCM]) as determined by core laboratory interpretation.
* Peak left ventricular outflow tract (LVOT) pressure gradient < 30 millimeters mercury (mm Hg) at rest and < 50 mm Hg with provocation (Valsalva maneuver and stress echocardiography).
* New York Heart Association (NYHA) Class II or III.

Exclusion Criteria

* Known infiltrative or storage disorder causing cardiac hypertrophy that mimics non-obstructive hypertrophic cardiomyopathy (nHCM) such as Fabry disease, amyloidosis, or Noonan syndrome with LV hypertrophy.
* History of unexplained syncope within 6 months prior to screening.
* History of sustained ventricular tachyarrhythmia (> 30 seconds) within 6 months prior to screening.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Kansas City Cardiomyopathy Questionnaire (23-item) Clinical Summary Score (KCCQ-23 CSS) at Week 48 | Up to Week 48
Change from baseline in peak oxygen consumption (pVO2) at Week 48 | Up to Week 48

SECONDARY OUTCOMES:
Change from baseline in ventilatory efficiency (VE/VCO2) slope to Week 48 | Up to Week 48
Proportion of participants with at least 1 class of New York Heart Association (NYHA) improvement from baseline to Week 48 | Up to Week 48
Change from baseline in N-terminal pro B-type natriuretic peptide (NT-proBNP) to Week 48 | Up to Week 48
Change from baseline in hypertrophic cardiomyopathy symptom questionnaire-shortness of breath (HCMSQ-SoB) domain to Week 48 | Up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (224):
- United States (41):
  - Local Institution - 0082, Birmingham, Alabama
  - Local Institution - 0458, Phoenix, Arizona
  - Local Institution - 0409, La Jolla, California
  - Local Institution - 0010, Los Angeles, California
  - Local Institution - 0406, San Francisco, California
  - Local Institution - 0079, Stanford, California
  - Local Institution - 0468, Gainesville, Florida
  - Local Institution - 0281, Tampa, Florida
  - Local Institution - 0092, Atlanta, Georgia
  - Local Institution - 0424, Indianapolis, Indiana
  - Local Institution - 0070, Iowa City, Iowa
  - Local Institution - 0410, Kansas City, Kansas
  - Local Institution - 0484, Louisville, Kentucky
  - Local Institution - 0127, Baltimore, Maryland
  - Local Institution - 0479, Boston, Massachusetts
  - Local Institution - 0500, Boston, Massachusetts
  - Local Institution - 0464, Ann Arbor, Michigan
  - Local Institution - 0064, Detroit, Michigan
  - Local Institution - 0455, Grand Rapids, Michigan
  - Local Institution - 0431, Rochester, Minnesota
  - Local Institution - 0461, St Louis, Missouri
  - Local Institution - 0435, Omaha, Nebraska
  - Local Institution - 0490, Morristown, New Jersey
  - Local Institution - 0449, Manhasset, New York
  - Local Institution - 0486, New York, New York
  - Local Institution - 0007, Stony Brook, New York
  - Local Institution - 0426, Valhalla, New York
  - Local Institution - 0094, Charlotte, North Carolina
  - Local Institution - 0065, Durham, North Carolina
  - Local Institution - 0083, Cleveland, Ohio
  - Local Institution - 0047, Hershey, Pennsylvania
  - Local Institution - 0444, Lancaster, Pennsylvania
  - Local Institution - 0263, Philadelphia, Pennsylvania
  - Local Institution - 0081, Pittsburgh, Pennsylvania
  - Local Institution - 0207, Germantown, Tennessee
  - Local Institution - 0089, Dallas, Texas
  - Local Institution - 0365, Dallas, Texas
  - Local Institution - 0492, Plano, Texas
  - Local Institution - 0402, Salt Lake City, Utah
  - Local Institution - 0478, Charlottesville, Virginia
  - Local Institution - 0095, Richmond, Virginia
- Australia (7):
  - Local Institution - 0063, Concord, New South Wales
  - Local Institution - 0085, Darlinghurst, New South Wales
  - Local Institution - 0369, Sydney, New South Wales
  - Local Institution - 0080, Chermside, Queensland
  - Local Institution - 0078, Milton, Queensland
  - Local Institution - 0050, Bedford Park, South Australia
  - Local Institution - 0076, Murdoch, Western Australia
- Austria (5):
  - Local Institution - 0090, Innsbruck, Tyrol
  - Local Institution - 0075, Linz, Upper Austria
  - Local Institution - 0069, Braunau am Inn, Upper Austria (Oberösterreich)
  - Local Institution - 0062, Graz
  - Local Institution - 0429, Vienna
- Belgium (4):
  - Local Institution - 0462, Edegem, Antwerpen
  - Local Institution - 0034, Anderlecht, Brussels Capital
  - Local Institution - 0476, Genk, Limburg
  - Local Institution - 0319, Leuven, Vlaams Brabant
- Brazil (11):
  - Local Institution - 0413, Salvador, Estado de Bahia
  - Local Institution - 0438, Brasília, Federal District
  - Local Institution - 0488, Belo Horizonte, Minas Gerais
  - Local Institution - 0447, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0450, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0430, Bragança Paulista, São Paulo
  - Local Institution - 0422, Ribeirão Preto, São Paulo
  - Local Institution - 0412, São Paulo, São Paulo
  - Local Institution - 0446, Rio de Janeiro
  - Local Institution - 0451, Rio de Janeiro
  - Local Institution - 0418, São Paulo
- Canada (5):
  - Local Institution - 0381, Calgary, Alberta
  - Local Institution - 0467, Vancouver, British Columbia
  - Local Institution - 0414, Hamilton, Ontario
  - Local Institution - 0411, London, Ontario
  - Local Institution - 0093, Québec, Quebec
- China (23):
  - Local Institution - 0535, Beijing, Beijing Municipality
  - Local Institution - 0534, Beijing, Beijing Municipality
  - Local Institution - 0503, Chongqing, Chongqing Municipality
  - Local Institution - 0541, Chongqing, Chongqing Municipality
  - Local Institution - 0539, Guangzhou, Guangdong
  - Local Institution - 0543, Guangzhou, Guangdong
  - Local Institution - 0549, Zhengzhou, Henan
  - Local Institution - 0542, Wuhan, Hubei
  - Local Institution - 0548, Changsha, Hunan
  - Local Institution - 0545, Suzhou, Jiangsu
  - Local Institution - 0550, Nanchang, Jiangxi
  - Local Institution - 0544, Changchun, Jilin
  - Local Institution - 0540, Dalian, Liaoning
  - Local Institution - 0501, Shenyang, Liaoning
  - Local Institution - 0538, Shenyang, Liaoning
  - Local Institution - 0547, Xi'an, Shan1xi
  - Local Institution - 0546, Jinan, Shandong
  - Local Institution - 0537, Shanghai, Shanghai Municipality
  - Local Institution - 0533, Chengdu, Sichuan
  - Local Institution - 0552, Chengdu, Sichuan
  - Local Institution - 0536, Wenzhou, Zhejiang
  - Local Institution - 0502, Beijing
  - Local Institution - 0553, Beijing
- Czechia (4):
  - Local Institution - 0086, Broumov, Královéhradecký kraj
  - Local Institution - 0052, Prague, Praha, Hlavní Mesto
  - Local Institution - 0033, Prague, Praha, Hlavní Mesto
  - Local Institution - 0188, Brno
- Denmark (3):
  - Local Institution - 0045, Aalborg, North Denmark
  - Local Institution - 0428, Aabenraa, Sønderjylland
  - Local Institution - 0019, Aarhus N
- France (11):
  - Local Institution - 0001, Nice, Alpes-Maritimes
  - Local Institution - 0463, Brest, Finistère
  - Local Institution - 0005, Toulouse, Haute-Garonne
  - Local Institution - 0003, Chambray-lès-Tours, Indre-et-Loire
  - Local Institution - 0489, La Tronche, Isère
  - Local Institution - 0067, Bron, Rhône
  - Local Institution - 0009, Nantes
  - Local Institution - 0004, Paris
  - Local Institution - 0006, Paris
  - Local Institution - 0053, Pessac
  - Local Institution - 0008, Rennes
- Germany (18):
  - Local Institution - 0404, Ulm, Baden-Wurttemberg
  - Local Institution - 0022, München, Bavaria
  - Local Institution - 0440, Regensburg, Bavaria
  - Local Institution - 0013, Bad Nauheim, Hesse
  - Local Institution - 0496, Göttingen, Lower Saxony
  - Local Institution - 0448, Hanover, Lower Saxony
  - Local Institution - 0273, Cologne, North Rhine Wesrphalia
  - Local Institution - 0439, Bad Oeynhausen, North Rhine-Westphalia
  - Local Institution - 0174, Bielefeld, North Rhine-Westphalia
  - Local Institution - 0420, Mainz, Rhineland-Palatinate
  - Local Institution - 0066, Lübeck, Schleswig-Holstein
  - Local Institution - 0016, Jena, Thuringia
  - Local Institution - 0403, Berlin
  - Local Institution - 0071, Freiburg im Breisgau
  - Local Institution - 0032, Hamburg
  - Local Institution - 0077, Heidelberg
  - Local Institution - 0454, München
  - Local Institution - 0046, Münster
- Hungary (5):
  - Local Institution - 0423, Balatonfüred, Veszprém megye
  - Local Institution - 0048, Budapest
  - Local Institution - 0039, Budapest
  - Local Institution - 0035, Budapest
  - Local Institution - 0417, Szeged
- India (5):
  - Local Institution - 0482, Ahmedabad, Gujarat
  - Local Institution - 0480, Bengaluru, Karnataka
  - Local Institution - 0481, Kochi, Kerala
  - Local Institution - 0483, Chandigarh
  - Local Institution - 0330, Gūrgaon
- Israel (9):
  - Local Institution - 0025, Jerusalem, Jerusalem
  - Local Institution - 0057, Jerusalem, Jerusalem
  - Local Institution - 0026, Ashkelon, Tel Aviv
  - Local Institution - 0037, Tel Aviv, Tel Aviv
  - Local Institution - 0419, Haifa
  - Local Institution - 0427, Petah Tikva
  - Local Institution - 0074, Ramat Gan
  - Local Institution - 0054, Rehovot
  - Local Institution - 0253, Safed
- Italy (3):
  - Local Institution - 0373, Florence, Tuscany
  - Local Institution - 0171, Pisa
  - Local Institution - 0028, Roma
- Japan (18):
  - Local Institution - 0370, Uwajima, Ehime
  - Local Institution - 0208, Himeji-Shi, Hyōgo
  - Local Institution - 0457, Kanazawa, Ishikawa-ken
  - Local Institution - 0107, Yokohama, Kanagawa
  - Local Institution - 0119, Nankoku-shi, Kochi
  - Local Institution - 0453, Tsu, Mie-ken
  - Local Institution - 0456, Sendai, Miyagi
  - Local Institution - 0452, Osaka, Osaka
  - Local Institution - 0315, Suita, Osaka
  - Local Institution - 0471, Takatsuki-Shi, Osaka
  - Local Institution - 0168, Hamamatsu, Shizuoka
  - Local Institution - 0477, Bunkyo-ku, Tokyo
  - Local Institution - 0505, Chuo-Ku, Tokyo
  - Local Institution - 0224, Itabashi-Ku, Tokyo
  - Local Institution - 0466, Koto-Ku, Tokyo
  - Local Institution - 0314, Shinjuku-ku, Tokyo
  - Local Institution - 0475, Shinjuku-ku, Tokyo
  - Local Institution - 0521, Fukuoka
- Netherlands (5):
  - Local Institution - 0442, Nijmegen, Gelderland
  - Local Institution - 0434, Maastricht, Limburg
  - Local Institution - 0197, Amsterdam-Zuidoost, North Holland
  - Local Institution - 0213, Rotterdam, South Holland
  - Local Institution - 0061, Utrecht
- Norway (3):
  - Local Institution - 0443, Lørenskog
  - Local Institution - 0441, Oslo
  - Local Institution - 0473, Trondheim
- Poland (11):
  - Local Institution - 0042, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0038, Wroclaw, Lower Silesian Voivodeship
  - Local Institution - 0091, Wroclaw, Lower Silesian Voivodeship
  - Local Institution - 0338, Warsaw, Masovian Voivodeship
  - Local Institution - 0203, Warsaw, Masovian Voivodeship
  - Local Institution - 0072, Rzeszów, Podkarpackie Voivodeship
  - Local Institution - 0017, Katowice, Silesian Voivodeship
  - Local Institution - 0415, Zabrze, Silesian Voivodeship
  - Local Institution - 0030, Bialystok
  - Local Institution - 0416, Lódz
  - Local Institution - 0059, Lodz, Łódź Voivodeship
- Portugal (6):
  - Local Institution - 0044, Guimarães, Braga District
  - Local Institution - 0015, Almada
  - Local Institution - 0433, Leiria
  - Local Institution - 0023, Lisbon
  - Local Institution - 0024, Lisbon
  - Local Institution - 0014, Vila Nova de Gaia
- South Korea (9):
  - Local Institution - 0516, Daegu, Daegu Gwang'yeogsi
  - Local Institution - 0518, Incheon, Incheon Gwang'yeogsi
  - Local Institution - 0012, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0055, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0460, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0517, Busan
  - Local Institution - 0508, Seongnam-si
  - Local Institution - 0217, Seoul
  - Local Institution - 0049, Seoul
- Spain (14):
  - Local Institution - 0040, Palma de Mallorca, Balearic Islands
  - Local Institution - 0299, L'Hospitalet de Llobregat, Barcelona
  - Local Institution - 0021, Majadahonda, Madrid
  - Local Institution - 0237, El Palmar, Murcia
  - Local Institution - 0043, A Coruña
  - Local Institution - 0087, Alicante
  - Local Institution - 0018, Barcelona
  - Local Institution - 0056, Barcelona
  - Local Institution - 0060, Granada
  - Local Institution - 0421, Madrid
  - Local Institution - 0041, Málaga
  - Local Institution - 0031, Salamanca
  - Local Institution - 0051, Seville
  - Local Institution - 0027, Valencia
- United Kingdom (4):
  - Local Institution - 0445, London, Greater London
  - Local Institution - 0073, Glasgow, Lanarkshire
  - Local Institution - 0407, Birmingham
  - Local Institution - 0472, London

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- [Derived] Desai MY, Owens AT, Abraham T, Olivotto I, Garcia-Pavia P, Lopes RD, Elliott P, Fernandes F, Verheyen N, Maier L, Meder B, Azevedo O, Kitaoka H, Wolski K, Wang Q, Jaber W, Mitchell L, Myers J, Rano T, Gong Z, Zhong Y, Carter-Bonanza S, Florea V, Aronson R, Nissen SE; ODYSSEY-HCM Investigators. Mavacamten in Symptomatic Nonobstructive Hypertrophic Cardiomyopathy. N Engl J Med. 2025 Sep 11;393(10):961-972. doi: 10.1056/NEJMoa2505927. Epub 2025 Aug 30. PMID 40888717
- [Derived] Desai MY, Olivotto I, Abraham T, Nissen SE, Garcia-Pavia P, Lopes RD, Elliott PM, Fernandes F, de Barros Correia E, Barriales-Villa R, Zorio E, Arad M, Shin SH, Verheyen N, Meder B, Azevedo O, Kitaoka H, Wolski K, Wang Q, Suryawanshi B, Wang Z, Florea V, Aronson R, Owens AT; ODYSSEY-HCM Investigators. Effects of Mavacamten on Cardiac Biomarkers in Nonobstructive Hypertrophic Cardiomyopathy: Insights From the ODYSSEY-HCM Trial. J Am Coll Cardiol. 2025 Dec 16;86(24):2418-2433. doi: 10.1016/j.jacc.2025.08.017. Epub 2025 Aug 27. PMID 40864018
- [Derived] Desai MY, Nissen SE, Abraham T, Olivotto I, Garcia-Pavia P, Lopes RD, Verheyen N, Wever-Pinzon O, Wolski K, Jaber W, Mitchell L, Davey D, Myers J, Rano T, Bhatia V, Zhong Y, Carter-Bonanza S, Florea V, Aronson R, Owens AT; ODYSSEY-HCM Investigators. Mavacamten in Symptomatic Nonobstructive Hypertrophic Cardiomyopathy: Design, Rationale, and Baseline Characteristics of ODYSSEY-HCM. JACC Heart Fail. 2025 Feb;13(2):358-370. doi: 10.1016/j.jchf.2024.11.013. PMID 39909647
- [Derived] O'Malley PA. Mavacamten (CAMZYOS) First-in-Class Small-Molecule Myosin Inhibitor for Treatment of Obstructive Hypertrophic Cardiomyopathy. Clin Nurse Spec. 2024 May-Jun 01;38(3):119-121. doi: 10.1097/NUR.0000000000000821. No abstract available. PMID 38625800
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com